CLINICAL TRIAL: NCT00548717
Title: Sirolimus, Mycophenolate Mofetil and Bortezomib as Graft-Versus-Host Disease Prophylaxis After Non-Myeloablative Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: Sirolimus, Mycophenolate Mofetil and Bortezomib as Graft-Versus-Host Disease (GVHD) Prophylaxis After Reduced Intensity Conditioning (RIC) Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: First two patients enrolled after trial reopened, developed grade III-IV acute GVHD and subsequently passed away.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); PDL BioPharma, Inc. (Industry)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DFCI 07-197
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Graft-vs-Host Disease
Keywords: GVHD; Stem cell transplantation; Sirolimus
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sirolimus; Mycophenolic Acid; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Siro/MMF (Experimental): Sirolimus and Mycophenolate Mofetil as GVHD Prophylaxis Sirolimus (Rapamycin); Mycophenolate Mofetil (MMF)
  Interventions: Drug: Sirolimus; Drug: Mycophenolate mofetil
- Siro/MMF/Bort (Experimental): Sirolimus, Mycophenolate Mofetil, and Bortezomib as GVHD Prophylaxis Sirolimus (Rapamycin); Mycophenolate Mofetil (MMF) Bortezomib (Velcade) *added with study reopening in 2012
  Interventions: Drug: Sirolimus; Drug: Mycophenolate mofetil; Drug: Bortezomib

INTERVENTIONS:
Drug: Sirolimus
  Other Names: Rapamycin
Drug: Mycophenolate mofetil
  Other Names: Cellcept
Drug: Bortezomib
  Other Names: Velcade
  Arms: Siro/MMF/Bort

SUMMARY:
This trial will test the hypothesis that the combination of sirolimus, mycophenolate mofetil, and bortezomib will be effective in preventing both acute and chronic GVHD after reduced intensity allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
The combination of tacrolimus and methotrexate is standard therapy for prevention of GVHD, however, our recent experience has demonstrated that the substitution of sirolimus for methotrexate provides superior GVHD control with reduced transplant-related toxicity. One limitation to the use of calcineurin inhibitors in GVHD prevention is the disruption in Treg function and proliferation. Based on our evolving understanding of the role of Treg in the development of chronic GVHD, we propose a GVHD prophylactic regimen that is effective in prevention of acute GVHD, but by virtue of the maintenance of Treg activity may be able to prevent chronic GVHD. We hypothesize that the substitution of mycophenolate mofetil for tacrolimus as well as the addition of bortezomib may provide similar protection against acute GVHD and prevent chronic GVHD while minimizing renal toxicity after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hematologic malignancies, who are at high risk of complications after conventional myeloablative transplantation
2. Patients must have a 6/6 matched, related donor. Matching at HLA Class II will be based on PCR of sequence specific primers (SSP). Among family member transplants, serologic matching at Class I is sufficient
3. Patient age greater than 18
4. Performance status 0-2
5. Life expectancy of > 100 days without transplantation
6. Written informed consent must be obtained in all cases from the patient

Exclusion Criteria:

1. Pregnancy
2. Prior Allogeneic Stem Cell Transplantation from any donor
3. Evidence of HIV infection or active Hepatitis B or C infection
4. Heart failure uncontrolled by medications
5. Total bilirubin > 2.0 mg/dl that is due to hepatocellular dysfunction
6. AST > 90
7. Cholesterol > 300 mg/dl or Triglycerides > 400 mg/dl while adequately treated
8. Uncontrolled bacterial, viral or fungal infection
9. Requirement for voriconazole at the time of hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Dana Farber Cancer Institute. The first participant was enrolled in November 2007. Enrollment was halted May 2008 due to an unacceptable rate of acute GVHD. The study reopened in November 2012 with addition of bortezomib. The last participant enrolled May 2013. The study was permanently closed to accural August 2013.
Groups:
- Siro/MMF: Sirolimus and Mycophenolate Mofetil as GVHD Prophylaxis
  Sirolimus (Rapamycin) Mycophenolate Mofetil (MMF)
- Siro/MMF/Bort: Sirolimus, Mycophenolate Mofetil, and Bortezomib for GVHD prophylaxis
  Sirolimus (Rapamycin) Mycophenolate Mofetil (MMF) Bortezomib (Velcade)
  *Bortezomib added when study reopened in November 2012
Period: Overall Study
Arm/Group | Siro/MMF | Siro/MMF/Bort
Started | 13 | 2
Completed | 4 | 0
Not Completed | 9 | 2
Not completed — Death | 5 | 2
Not completed — Relapse | 3 | 0
Not completed — Alternative treatment for GVHD | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Siro/MMF: Sirolimus and Mycophenolate Mofetil as GVHD Prophylaxis
  Sirolimus (Rapamycin); Mycophenolate Mofetil (MMF);
- Siro/MMF/Bort: Sirolimus, Mycophenolate Mofetil, and Bortezomib as GVHD Prophylaxis
  Sirolimus (Rapamycin); Mycophenolate Mofetil (MMF); Bortezomib (Velcade) *added with study reopening in 2012
- Total: Total of all reporting groups
Arm/Group | Siro/MMF | Siro/MMF/Bort | Total
Number analyzed (Participants) | 13 | 2 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 0 | 11
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 9 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 13 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Rate of Grade II-IV Acute GVHD When Sirolimus and Mycophenolate Mofetil or Sirolimus, Mycophenolate Mofetil and Bortezomib is Used for GVHD Prophylaxis After Allogeneic Stem Cell Transplantation in Patients With Hematologic Malignancies
Time Frame: 150 days
Measure: Number; unit: percentage of participants
Groups:
- Siro/MMF/Bort: Sirolimus, Mycophenolate Mofetil, and Bortezomib as GVHD Prophylaxis
  Sirolimus (Rapamycin); Mycophenolate Mofetil (MMF);Bortezomib (Velcade) *added with study reopening in 2012
Arm/Group | Siro/MMF | Siro/MMF/Bort
Number analyzed (Participants) | 13 | 2
percentage of participants | 77 | 100

2. Secondary Outcome: Donor Stem Cell Engraftment, Including Donor-host Hematopoietic Chimerism Studies Post Transplant
Description: Engraftment of donor cells by week 4 after transplantation. Assessment of donor stem cell engraftment will include donor-host hematopoietic chimerism analyses at 4 weeks and every 3 months after transplantation. Chimerism measured from peripheral blood or from bone marrow.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Siro/MMF | Siro/MMF/Bort
Number analyzed (Participants) | 13 | 2
participants | 9 | 2

3. Secondary Outcome: The Rate of Renal Insufficiency
Description: Renal function will be measured weekly after transplant for 4 weeks, at 8 weeks and then at 3 month intervals from transplantation. Sentinel renal events such as the occurrence of thrombotic microangiopathy will be noted.
  The rationale for the substitution of mycophenolate mofetil for tacrolimus is to continue to prevent acute GVHD, but minimize renal toxicity after transplantation. We will thus monitor renal toxicity closely in this study. In our previous experience, the rate of grade III-V renal toxicity by day 100 after transplantation was about 10%. Here, grade III is defined as a creatinine level between 3.1 to 6 times the normal level, grade IV is defined as a creatinine level 6 times or more the normal level, and grade V is defined as a fatality due to renal toxicity.
Time Frame: 1 year
Population: One patient experienced grade 5 renal toxicity
Measure: Number; unit: participants
Arm/Group | Siro/MMF | Siro/MMF/Bort
Number analyzed (Participants) | 13 | 2
participants | 1 | 0

4. Secondary Outcome: To Correlate the Serum Concentrations of Mycophenolate Mofetil and Its Metabolites With Acute GVHD Incidence
Description: This outcome measure was presented as a comparison between incidence of Grade 0-I aGVHD and Grade II-IV aGVHD across 5 time points (Weeks 1,2,3,8, and 12).
Time Frame: 1 year
Population: In the Siro/MMF group, the overall number of participants analyzed was 13, however, the number of participants with the MMF level data available varies at each time point. For the Siro/MMF/Bort group, no data were analyzed due to no data available for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Siro/MMF | Siro/MMF/Bort
Number analyzed (Participants) | 13 | 0
ng/mL
  Week 1 MMF level (0-I aGVHD), n=3 | 2.43 (1.19) |
  Week 1 MMF level (II-IV aGVHD), n=8 | 2.70 (1.25) |
  Week 2 MMF level (0-I aGVHD), n=3 | 3.40 (1.37) |
  Week 2 MMF level (II-IV aGVHD), n=6 | 3.07 (2.25) |
  Week 3 MMF level (0-I aGVHD), n=3 | 2.57 (1.35) |
  Week 3 MMF level (II-IV aGVHD), n=6 | 2.85 (2.09) |
  Week 8 MMF level (0-I aGVHD), n=3 | 2.37 (0.75) |
  Week 8 MMF level (II-IV aGVHD), n=4 | 2.13 (1.18) |
  Week 12 MMF level (0-I aGVHD), n=2 | 1.75 (0.07) |
  Week 12 MMF level (II-IV aGVHD), n=4 | 2.20 (1.19) |
Statistical Analysis 1: Comparison: Siro/MMF; Comparison between Grade 0-I aGVHD vs Grade II-IV aGVHD in the Siro/MMF group at week 1; Test type: Superiority or Other; p = 0.77, t-test, 2 sided
Statistical Analysis 2: Comparison: Siro/MMF; Comparison between Grade 0-I aGVHD vs Grade II-IV aGVHD in the Siro/MMF group at week 2; Test type: Superiority or Other; p = 0.59, t-test, 2 sided
Statistical Analysis 3: Comparison: Siro/MMF; Comparison between Grade 0-I aGVHD vs Grade II-IV aGVHD in the Siro/MMF group at week 3; Test type: Superiority or Other; p = 0.92, t-test, 2 sided
Statistical Analysis 4: Comparison: Siro/MMF; Comparison between Grade 0-I aGVHD vs Grade II-IV aGVHD in the Siro/MMF group at week 8; Test type: Superiority or Other; p = 0.63, t-test, 2 sided
Statistical Analysis 5: Comparison: Siro/MMF; Comparison between Grade 0-I aGVHD vs Grade II-IV aGVHD in the Siro/MMF group at week 12; Test type: Superiority or Other; p = 0.79, t-test, 2 sided

5. Secondary Outcome: Incidence of 100 Day Mortality
Time Frame: 100 days
Measure: Number; unit: percentage of participants
Arm/Group | Siro/MMF | Siro/MMF/Bort
Number analyzed (Participants) | 13 | 2
percentage of participants | 31 | 0

6. Secondary Outcome: Incidence of Chronic GVHD
Description: Chronic GVHD will be graded according to the modified Seattle criteria. Chronic GVHD divided into limited and extensive and evaluated across the following systems: skin, cutaneous structures, liver, mouth, eyes, esophagus, intestines, lung, musculoskeletal, serous, nervous, urologic, vagina, hematopoietic, and immune.
  Localized skin involvement with or without hepatic dysfunction is classified as limited disease.
  Generalized skin involvement or limited disease plus eye involvement, oral involvement, hepatic dysfunction with abnormal liver histology, or involvement of any other target organ was classified as extensive disease.
  Lee SJ, Vogelsang G, Flowers ME. Chronic graft-versus-host disease. Biol Blood Marrow Transplant.
  2003;9:215-33.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Groups:
- Siro /MMF: Sirolimus and Mycophenolate Mofetil as GVHD Prophylaxis
  Sirolimus (Rapamycin); Mycophenolate Mofetil (MMF);
- Siro/MMF/Bort: Sirolimus, Mycophenolate Mofetil,and Bortezomib as GVHD Prophylaxis
  Sirolimus (Rapamycin); Mycophenolate Mofetil (MMF); Bortezomib (Velcade) *added with study reopening in 2012
Arm/Group | Siro /MMF | Siro/MMF/Bort
Number analyzed (Participants) | 13 | 2
percentage of participants | 15 | 50

7. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Siro/MMF | Siro/MMF/Bort
Number analyzed (Participants) | 13 | 2
percentage of participants | 39 | 0

ADVERSE EVENTS:
Time Frame: Participating investigators will assess the occurrence of AEs and SAEs at all participant evaluation time points during the study. All SAEs and grade 3 or higher treatment and/or transplant related toxicities (AEs) are recorded.
Description: It is not simple to segregate prophylactic regimen related from transplant related toxicities. We thus report transplant and/or regimen related toxicities combined and do not segregate toxicities by regimen. Moreover, since only 2 patients received Siro/MMF/Bort, comparison of toxicites between the two regimens is infeasible.
Groups:
- Siro/MMF (+/- Bortezomib): Sirolimus and Mycophenolate Mofetil as GVHD Prophylaxis (+/- Bortezomib)
  Sirolimus (Rapamycin); Mycophenolate Mofetil (MMF); Bortezomib (Velcade) *added with study reopening in 2012
Arm/Group | Siro/MMF (+/- Bortezomib)
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Siro/MMF (+/- Bortezomib) (N=15)
Fever (General disorders) | 1 (1)
Multi-organ Failure (General disorders) | 1 (1)
GVHD (Immune system disorders) | 2 (2)
HHV6 encephalitis (Infections and infestations) | 1 (1)
Temporary blindness (Eye disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siro/MMF (+/- Bortezomib) (N=15)
Documented infection (Infections and infestations) | 7
Suspected Undocumented infection (Infections and infestations) | 4
Cholecystitis (Hepatobiliary disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1 — w/o prior colostomy
Encephalopathy (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Necrosis-small bowel NOS (Gastrointestinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Renal Toxicity (Renal and urinary disorders) | 1
Neurologic Toxicity (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Results are reported for transparency only, and should not be used to extrapolate significant conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes